CLINICAL TRIAL: NCT03743571
Title: Augmenting Exposure Therapy for Social Anxiety With Transcranial Direct Current Stimulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment terminated due to COVID-related social distancing requirements
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1222479-2
Record Dates: First submitted 2018-11-09; First posted 2018-11-16 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-08

CONDITIONS: Social Anxiety
Keywords: social anxiety; transcranial direct current stimulation; exposure therapy
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Implosive Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either sham or anodal (2 mA) tDCS targeting the mPFC during exposure therapy for public speaking anxiety.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- anodal tDCS during exposure (Active Comparator): anodal transcranial direct current stimulation (2mA) will be applied over EEG coordinate FpZ to target mPFC activation during exposure therapy
  Interventions: Device: transcranial direct current stimulation; Behavioral: exposure therapy
- sham tDCS during exposure (Sham Comparator): sham transcranial direct current stimulation will be applied over EEG coordinate FpZ during exposure therapy at a level that provides the physical sensations of tDCS but which is non-therapeutic
  Interventions: Device: transcranial direct current stimulation; Behavioral: exposure therapy

INTERVENTIONS:
Device: transcranial direct current stimulation — tDCS will be applied over EEG coordinate FpZ to target mPFC activation during exposure therapy
Behavioral: exposure therapy — participants will complete one session of exposure therapy for fear of public speaking, which will involve providing speeches to audiences in virtual reality

SUMMARY:
This study will examine whether transcranial direct current stimulation (tDCS) can be used to improve outcomes from exposure therapy for social anxiety disorder, and facilitate extinction of fear responding toward individuals outside one's own ethnic group (i.e., ethnic out-group members).

DETAILED DESCRIPTION:
Although exposure therapy is among the most powerful treatment techniques for social anxiety, many individuals do not achieve full remission. Furthermore, some research suggests that fear responding toward ethnic out-group members may be more resistant to extinction. Enhancing activation of the mPFC during exposure therapy may improve overall response to treatment, and also facilitate extinction of fear toward ethic out-groups. Researchers have found that greater mPFC activation during exposure therapy is associated with better outcomes, and that transcranial direct current stimulation (tDCS) can be used enhance learning and cognition with no known serious adverse effects. This study will therefore examine whether active/anodal (versus sham) tDCS targeting the mPFC (a) enhances overall reductions in social anxiety symptoms, and (b) facilitates extinction of fear responding toward ethnic/racial out-groups for both Latino and Caucasian/non-Latino participants. Participants will receive either active/anodal tDCS or sham tDCS during a brief exposure therapy intervention involving public speaking in a Virtual Reality (VR) environment. The public speaking audience in the VR environment will alternate between audiences that are either matched or unmatched to the participant's ethnicity (in a randomly assigned order). Participants' fear reactivity will be assessed with behavioral, physiological, and subjective measures at baseline, post-treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older (adult)
* Enrolled in higher education (post-high school)
* Elevated public speaking anxiety as indicated by self-report questions
* NOT currently receiving in exposure therapy for social anxiety

Exclusion Criteria:

* History of seizure or any other neurological diagnosis
* Has any metal in their skull (plates, steel sutures, etc.)
* Participant is currently taking anti-convulsant, sedative/hypnotic, or antipsychotic medications
* Participant is pregnant
* Participant has already participated in a prior tDCS/tACS study on the same day as study visit 1 (which will involve either placebo or active/anodal tDCS stimulation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada, Reno, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
Study protocols and de-identified data will be shared at the request of other researchers.

REFERENCES:
- [Result] McDonald MA, Meckes SJ, Shires J, Berryhill ME, Lancaster CL. Augmenting Virtual Reality Exposure Therapy for Social and Intergroup Anxiety With Transcranial Direct Current Stimulation. J ECT. 2024 Mar 1;40(1):51-60. doi: 10.1097/YCT.0000000000000967. Epub 2023 Nov 24. PMID 38009966

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anodal tDCS During Exposure | Sham tDCS During Exposure
Started | 17 | 16
Completed | 15 | 13
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Population: Participants who withdrew from the study (n = 2) were not included in the baseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anodal tDCS During Exposure | Sham tDCS During Exposure | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.75 (1.45) | 20 (1.51) | 19.87 (1.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 20
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 13 | 26
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 15 | 31
BAT: Matched Audience, Speech Duration [Mean (Standard Deviation); unit: seconds] — During Behavioral Approach Tests (BATs), participants will provide a speech to (a) an audience primarily matched to their ethnicity, and (b) an audience primarily un-matched to their ethnicity. The speech will be for up to 5 minutes in duration. During each BAT, we will assess fear response behaviorally (length of the speech, up to 5 min in duration) and subjectively (self reported levels of anticipated and peak fear). ***This report is for the baseline duration of the matched BAT. The range is from 0 to 300 seconds. Longer speech durations indicate greater approach, and a better outcome.***
  seconds | 112 (49) | 159 (94) | 135 (76)
BAT: Matched Audience, Anticipated Anxiety [Mean (Standard Deviation); unit: units on a scale] — During Behavioral Approach Tests (BATs), participants provide a speech to (a) an audience primarily matched to their ethnicity, and (b) an audience primarily un-matched to their ethnicity. The speech will be for up to 5 minutes in duration. During each BAT, we will assess fear response behaviorally (length of the speech, up to 5 min in duration) and subjectively (self reported levels of anticipated and peak anxiety). **This report is for the baseline anticipated anxiety rating for the matched BAT. The range of the subjective rating is 0 to 100, with higher scores indicating a worse outcome.** Population: Anticipated anxiety ratings at baseline (BAT matched and unmatched) were missing for one participant in the anodal tDCS condition (n= 15 total, instead of n = 16 for this measure only), due to an experimenter error.
  units on a scale
    number analyzed (Participants) | 15 | 15 | 30
    (all) | 70 (16) | 64 (29) | 67 (23)
BAT: Matched Audience, Peak Anxiety [Mean (Standard Deviation); unit: units on a scale] — During Behavioral Approach Tests (BATs), participants provide a speech to (a) an audience primarily matched to their ethnicity, and (b) an audience primarily un-matched to their ethnicity. The speech will be for up to 5 minutes in duration. During each BAT, we will assess fear response behaviorally (length of the speech, up to 5 min in duration) and subjectively (self reported levels of anticipated and peak anxiety). ***This report is for the baseline peak anxiety rating for the matched BAT. The range of the subjective rating is 0 to 100, with higher scores indicating a worse outcome.***
  units on a scale | 59 (31) | 65 (24) | 62 (27)
BAT: Unmatched Audience, Speech Duration [Mean (Standard Deviation); unit: units on a scale] — During Behavioral Approach Tests (BATs), participants will provide a speech to (a) an audience primarily matched to their ethnicity, and (b) an audience primarily un-matched to their ethnicity. The speech will be for up to 5 minutes in duration. During each BAT, we will assess fear response behaviorally (length of the speech, up to 5 min in duration) and subjectively (self reported levels of anticipated and peak fear). ***This report is for the baseline duration of the unmatched BAT. The range is from 0 to 300 seconds. Longer speech durations indicate greater approach, and a better outcome.***
  units on a scale | 121 (75) | 155 (103) | 137 (90)
BAT: Unmatched Audience, Anticipated Anxiety [Mean (Standard Deviation); unit: units on a scale] — During Behavioral Approach Tests (BATs), participants provide a speech to (a) an audience primarily matched to their ethnicity, and (b) an audience primarily un-matched to their ethnicity. The speech will be for up to 5 minutes in duration. During each BAT, we will assess fear response behaviorally (length of the speech, up to 5 min in duration) and subjectively (self reported levels of anticipated and peak anxiety). *This report is for the baseline anticipated anxiety rating for the unmatched BAT. The range of the subjective rating is 0 to 100, with higher scores indicating a worse outcome.* Population: Anticipated anxiety ratings at baseline (BAT matched and unmatched) were missing for one participant in the anodal tDCS condition (n= 15 total, instead of n = 16 for this measure only), due to an experimenter error.
  units on a scale
    number analyzed (Participants) | 15 | 15 | 30
    (all) | 66 (22) | 69 (22) | 68 (22)
BAT: Unmatched Audience, Peak Anxiety [Mean (Standard Deviation); unit: units on a scale] — During Behavioral Approach Tests (BATs), participants provide a speech to (a) an audience primarily matched to their ethnicity, and (b) an audience primarily un-matched to their ethnicity. The speech will be for up to 5 minutes in duration. During each BAT, we will assess fear response behaviorally (length of the speech, up to 5 min in duration) and subjectively (self reported levels of anticipated and peak anxiety). ***This report is for the baseline peak anxiety rating for the unmatched BAT. The range of the subjective rating is 0 to 100, with higher scores indicating a worse outcome.***
  units on a scale | 69 (27) | 72 (21) | 71 (24)
Personal Report of Public Speaking Anxiety [Mean (Standard Deviation); unit: units on a scale] — Participants will complete the Personal Report of Public Speaking Anxiety (PRPSA), a 34-item questionnaire that assesses public speaking anxiety. The items are sum scored, and totals range from 34 to 170, with higher scores indicating a worse outcome.
  units on a scale | 149 (9) | 145 (11) | 147 (10)
Positive Self Statements [Mean (Standard Deviation); unit: units on a scale] — Participants will complete the Positive Self Statements subscale of the Self Statements During Public Speaking Scale (SSPS). The SSPS is 10-item questionnaire that asses both positive and negative self statements associated with public speaking. The items within each of the two subscales are summed, with total scores ranging from 0 to 25 for each subscale, and higher scores indicating higher levels of agreement with positive or negative self statements, respectively. Higher scores on the positive self statements indicate a better outcome.
  units on a scale | 10 (3) | 10 (4) | 10 (4)
Negative Self Statements [Mean (Standard Deviation); unit: units on a scale] — Participants will complete the Negative Self Statements subscale of the Self Statements During Public Speaking Scale (SSPS). The SSPS is 10-item questionnaire that asses both positive and negative self statements associated with public speaking. The items within each of the two subscales are summed, with total scores ranging from 0 to 25 for each subscale, and higher scores indicating higher levels of agreement with positive or negative self statements, respectively. Higher scores on the negative self statements indicate a worse outcome.
  units on a scale | 14 (3) | 13 (4) | 14 (4)

OUTCOME MEASURES:

1. Primary Outcome: BAT: Matched Audience, Speech Duration
Description: During Behavioral Approach Tests (BATs), participants will provide a speech to (a) an audience primarily matched to their ethnicity, and (b) an audience primarily un-matched to their ethnicity. The speech will be for up to 5 minutes in duration. During each BAT, we will assess fear response behaviorally (length of the speech, up to 5 min in duration) and subjectively (self reported levels of anticipated and peak fear).
  ***This outcome report is for the duration of the matched BAT. The total possible range of the speech is from 0 to 300 seconds. Longer speech durations indicate greater approach, which is a better outcome.***
Time Frame: follow-up, one month after baseline assessment
Population: Completer-only analysis (no imputation).
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Anodal tDCS During Exposure | Sham tDCS During Exposure
Number analyzed (Participants) | 14 | 12
seconds | 129 (52) | 141 (65)
Statistical Analysis 1: Comparison: Anodal tDCS During Exposure vs Sham tDCS During Exposure; We used a null hypothesis significance testing approach in our analyses. For performance on Behavioral Approach Tests (BATs), we completed 2 x 2 x 2 mixed factorial ANOVAs to evaluate the impact of tDCS groups (between-subjects variable; anodal/active vs sham), time (within subjects variable; baseline vs follow-up), and audience type (ethnicity primary matched vs unmatched to the participants' own identity) on outcome measures; Test type: Other — We needed a total sample size of at least N = 24 to reach 80% power to detect a moderately large effect (Cohen's f = 0.3) for 2x2 interactions to determine whether scores differed across time (baseline vs follow up) for the two tDCS groups (anodal/active vs sham), and whether scores differed between audience type (matched vs unmatched) for the two tDCS groups (anodal/active vs sham); p = .42, ANOVA — Unadjusted. A priori threshold was set at p < .05, two-tailed; tDCS (anodal vs sham) x Time (baseline vs follow-up) interaction: F(1,24) = 0.67, p = 0.42

2. Primary Outcome: BAT: Matched Audience, Anticipated Anxiety
Description: During Behavioral Approach Tests (BATs), participants will provide a speech to (a) an audience primarily matched to their ethnicity, and (b) an audience primarily un-matched to their ethnicity. The speech will be for up to 5 minutes in duration. During each BAT, we will assess fear response behaviorally (length of the speech, up to 5 min in duration) and subjectively (self reported levels of anticipated and peak anxiety).
  ***This outcome report is for anticipated anxiety during the matched BAT. The total possible range of the subjective rating is from 0 to 100. Higher ratings indicate greater anxiety, which is a worse outcome.***
Time Frame: follow-up, one month after baseline assessment
Population: Completer only (no imputation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anodal tDCS During Exposure | Sham tDCS During Exposure
Number analyzed (Participants) | 14 | 12
units on a scale | 39 (19) | 38 (25)
Statistical Analysis 1: Comparison: Anodal tDCS During Exposure vs Sham tDCS During Exposure; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .88, ANOVA — Unadjusted. A priori threshold was set at p < .05, two-tailed; tDCS (anodal vs sham) x Time (baseline vs follow-up) interaction: F(1,24) = 0.02, p = .88

3. Primary Outcome: BAT: Matched Audience, Peak Anxiety
Description: During Behavioral Approach Tests (BATs), participants will provide a speech to (a) an audience primarily matched to their ethnicity, and (b) an audience primarily un-matched to their ethnicity. The speech will be for up to 5 minutes in duration. During each BAT, we will assess fear response behaviorally (length of the speech, up to 5 min in duration) and subjectively (self reported levels of anticipated and peak anxiety).
  ***This outcome report is for peak anxiety during the matched BAT. The total possible range of the subjective rating is from 0 to 100. Higher ratings indicate greater anxiety, which is a worse outcome.***
Time Frame: follow-up, one month after baseline assessment
Population: completers only (no imputation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anodal tDCS During Exposure | Sham tDCS During Exposure
Number analyzed (Participants) | 14 | 12
units on a scale | 36 (21) | 26 (27)
Statistical Analysis 1: Comparison: Anodal tDCS During Exposure vs Sham tDCS During Exposure; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .17, ANOVA — Unadjusted. A priori threshold was set at p < .05, two-tailed; tDCS (anodal vs sham) x Time (baseline vs follow-up) interaction: F(1,24) = 1.98, p = .17

4. Primary Outcome: BAT: Unmatched Audience, Speech Duration
Description: During Behavioral Approach Tests (BATs), participants will provide a speech to (a) an audience primarily matched to their ethnicity, and (b) an audience primarily un-matched to their ethnicity. The speech will be for up to 5 minutes in duration. During each BAT, we will assess fear response behaviorally (length of the speech, up to 5 min in duration) and subjectively (self reported levels of anticipated and peak fear).
  ***This outcome report is for the duration of the unmatched BAT. The total possible range of the speech is from 0 to 300 seconds. Longer speech durations indicate greater approach, which is a better outcome.***
Time Frame: follow-up, one month after baseline assessment
Population: completers only (no imputation).
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Anodal tDCS During Exposure | Sham tDCS During Exposure
Number analyzed (Participants) | 14 | 12
seconds | 145 (60) | 168 (72)
Statistical Analysis 1: Comparison: Anodal tDCS During Exposure vs Sham tDCS During Exposure; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .42, ANOVA — Unadjusted. A priori threshold was set at p < .05, two-tailed; tDCS (anodal vs sham) x Time (baseline vs follow-up) interaction: F(1,24) = 0.67, p = 0.42

5. Primary Outcome: BAT: Unmatched Audience, Anticipated Anxiety
Description: During Behavioral Approach Tests (BATs), participants will provide a speech to (a) an audience primarily matched to their ethnicity, and (b) an audience primarily un-matched to their ethnicity. The speech will be for up to 5 minutes in duration. During each BAT, we will assess fear response behaviorally (length of the speech, up to 5 min in duration) and subjectively (self reported levels of anticipated and peak anxiety).
  ***This outcome report is for anticipated anxiety during the unmatched BAT. The total possible range of the subjective rating is from 0 to 100. Higher ratings indicate greater anxiety, which is a worse outcome.***
Time Frame: follow-up, one month after baseline assessment
Population: completers only (no imputation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anodal tDCS During Exposure | Sham tDCS During Exposure
Number analyzed (Participants) | 14 | 12
units on a scale | 43 (21) | 40 (25)
Statistical Analysis 1: Comparison: Anodal tDCS During Exposure vs Sham tDCS During Exposure; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .88, ANOVA — Unadjusted. A priori threshold was set at p < .05, two-tailed; tDCS (anodal vs sham) x Time (baseline vs follow-up) interaction: F(1,24) = 0.02, p = .88

6. Primary Outcome: BAT: Unmatched Audience, Peak Anxiety
Description: During Behavioral Approach Tests (BATs), participants will provide a speech to (a) an audience primarily matched to their ethnicity, and (b) an audience primarily un-matched to their ethnicity. The speech will be for up to 5 minutes in duration. During each BAT, we will assess fear response behaviorally (length of the speech, up to 5 min in duration) and subjectively (self reported levels of anticipated and peak anxiety).
  ***This outcome report is for peak anxiety during the unmatched BAT. The total possible range of the subjective rating is from 0 to 100. Higher ratings indicate greater anxiety, which is a worse outcome.***
Time Frame: follow-up, one month after baseline assessment
Population: completers only (no imputation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anodal tDCS During Exposure | Sham tDCS During Exposure
Number analyzed (Participants) | 14 | 12
units on a scale | 35 (21) | 28 (24)
Statistical Analysis 1: Comparison: Anodal tDCS During Exposure vs Sham tDCS During Exposure; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .17, ANOVA — Unadjusted. A priori threshold was set at p < .05, two-tailed; tDCS (anodal vs sham) x Time (baseline vs follow-up) interaction: F(1,24) = 1.98, p = .17

7. Secondary Outcome: Personal Report of Public Speaking Anxiety
Description: Participants will complete the Personal Report of Public Speaking Anxiety (PRPSA), a 34-item questionnaire that assesses public speaking anxiety. The items are sum scored, and totals range from 34 to 170, with higher scores indicating higher levels of public speaking anxiety.
Time Frame: follow-up, one month after baseline assessment
Population: completer only (no imputation). Note: Three additional participants were excluded from the primary outcome data, but not secondary outcome data. Social distancing guidelines prevented them from attending a lab visit to complete the primary outcome measure (the BATs), but they were able to complete the secondary outcome measures remotely (questionnaires).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anodal tDCS During Exposure | Sham tDCS During Exposure
Number analyzed (Participants) | 15 | 13
score on a scale | 133.47 (16.69) | 131.15 (17.87)
Statistical Analysis 1: Comparison: Anodal tDCS During Exposure vs Sham tDCS During Exposure; We used a null hypothesis significance testing approach in our analyses. For performance on the questionnaires, we completed 2 x 2 mixed factorial ANOVAs to evaluate the impact of tDCS groups (between-subjects variable; anodal/active vs sham) and time (within subjects variable; baseline vs follow-up) on outcome measures; Test type: Other — We needed a total sample size of at least N = 24 to reach 80% power to detect a moderately large effect (Cohen's f = 0.3) for 2x2 interactions to determine whether scores differed across time (baseline vs follow up) for the two tDCS groups (anodal/active vs sham); p = .67, ANOVA — Unadjusted. A priori threshold was set at p < .05, two-tailed; tDCS (anodal vs sham) x Time (baseline vs follow-up) interaction: F(1,26) = 0.19, p = .67

8. Secondary Outcome: Positive Self Statements
Description: Participants will complete the Positive Self Statements subscale of the Self Statements During Public Speaking Scale (SSPS). The SSPS is 10-item questionnaire that asses both positive and negative self statements associated with public speaking. The items within each of the two subscales are summed, with total scores ranging from 0 to 25 for each subscale, and higher scores indicating higher levels of agreement with positive or negative self statements, respectively. Higher scores on the positive self statements indicate less anxiety.
Time Frame: follow-up, one month after baseline assessment
Population: completers only (no imputation). Note: Three additional participants were excluded from the primary outcome data, but not secondary outcome data. Social distancing guidelines prevented them from attending a lab visit to complete the primary outcome measure (the BATs), but they were able to complete the secondary outcome measures remotely (questionnaires).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anodal tDCS During Exposure | Sham tDCS During Exposure
Number analyzed (Participants) | 15 | 13
score on a scale | 11.13 (5.14) | 10.69 (4.57)
Statistical Analysis 1: Comparison: Anodal tDCS During Exposure vs Sham tDCS During Exposure; [analysis description as in outcome 7, analysis 1]; Test type: Other — [test comment as in outcome 7, analysis 1]; p = .96, ANOVA — Unadjusted. A priori threshold was set at p < .05, two-tailed; tDCS (anodal vs sham) x Time (baseline vs follow-up) interaction: F(1,26) < .01, p = .96

9. Secondary Outcome: Negative Self Statements
Description: Participants will complete the Negative Self Statements subscale of the Self Statements During Public Speaking Scale (SSPS). The SSPS is 10-item questionnaire that asses both positive and negative self statements associated with public speaking. The items within each of the two subscales are summed, with total scores ranging from 0 to 25 for each subscale, and higher scores indicating higher levels of agreement with positive or negative self statements, respectively. Higher scores on the negative self statements indicate more anxiety.
Time Frame: follow-up, one month after baseline assessment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anodal tDCS During Exposure | Sham tDCS During Exposure
Number analyzed (Participants) | 15 | 13
score on a scale | 12.33 (6.95) | 11.77 (6.83)
Statistical Analysis 1: Comparison: Anodal tDCS During Exposure vs Sham tDCS During Exposure; [analysis description as in outcome 7, analysis 1]; Test type: Other — We needed a total sample size of at least N = 24 to reach 80% power to detect a moderately large effect (Cohen's f = 0.3) for 2x2 interactions to determine whether scores differed across time (baseline vs follow up) for the two tDCS groups (anodal/active vs sham),; p = .43, ANOVA — Unadjusted. A priori threshold was set at p < .05, two-tailed; tDCS (anodal vs sham) x Time (baseline vs follow-up) interaction: F(1,26) = 0.65, p = .43

ADVERSE EVENTS:
Time Frame: The timeframe for data collection for the project. This included baseline (enrollment day) through follow-up, which was approximately one month after enrollment.
Description: Definitions were consistent with clinicaltrials.gov
Arm/Group | Anodal tDCS During Exposure | Sham tDCS During Exposure
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT03743571/Prot_SAP_000.pdf